CLINICAL TRIAL: NCT02074176
Title: Plasma Orexin A and mRNA Expression Levels of Pre-pro-orexin Gene in Attention-Deficit Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201008049R
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Attention-deficit/hyperactivity disorder; orexin A; mRNA
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — mRNA,pre-pro-orexin gene
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: Attention deficit hyperactivity disorder (ADHD) is an early onset, highly heritable, clinically heterogeneous, long-term impairing disorder with tremendous impact on individuals, families, and societies. It affects 7.5% of school-aged children in Taiwan. Emerging evidence has suggested that patients with ADHD may present with a deficit of attention, alertness and sleep disturbances. Since attention, alertness, and sleep disturbances may significantly increase the functional impairment of ADHD, gaining insight into their pathophysiology as well as into their treatment is of relevance to provide a better clinical management of patients suffering from ADHD. The orexin system, located in the hypothalamus, takes an important role in homeostatic functions, such as attention, alertness, sleep-wake cycle, and feeding. To our best knowledge, the functioning of the orexin system has never been investigated in patients with ADHD. Given the involvement of the orexin system in the control of alertness and reward seeking, the present study aims to examine whether plasma orexin and mRNA expression levels of pre-pro-orexin gene are associated with the symptoms and neurocognitive deficits of ADHD.

DETAILED DESCRIPTION:
Specific Aims:

1. To evaluate the correlations between plasma levels of orexin A and symptoms of ADHD.
2. To evaluate the correlations between mRNA expression levels of pre-pro-orexin gene and symptoms of ADHD.
3. To evaluate the correlations between plasma levels of orexin A and neurocognitive dysfunction of ADHD.
4. To evaluate the correlations between mRNA expression levels of pre-pro-orexin gene and neurocognitive dysfunction of ADHD.

Subjects and Methods: Subjects in this study will be recruited from Children's Mental Health Center, Department of Psychiatry, National Taiwan University Hospital (NTUH). The sample will consist of 50 ADHD probands (aged 6 to 18 years) and 50 age- and sex- matched healthy controls. The phenotype measures include (1) interviews for psychopathology (K-SADS-E) and social functioning (SAICA), (2) self-administered questionnaires to measures ADHD symptoms (SNAP-IV), comorbid conditions (YSR, CBCL), and family support (Family APGAR), and (3) Neuropsychological tests: CPT, WISC-III, and CANTAB. Plasma orexin A and mRNA expression levels of pre-pro-orexin gene will be measured in all participants.

Anticipated Results: We anticipate the identification of potential relationship between plasma orexin A, mRNA expression and symptoms of ADHD. In addition, this study will determine the association of plasma orexin A and mRNA expression with the neurocognitive deficits of ADHD. We hope that this study will elucidate the pathogenesis of ADHD, and orexin A will be a possible biomarker for this disorder. In addition, the data of orexin A and mRNA expression of pre-pro-orexin gene in ADHD will provide insight in developing more specific and more effective treatment for ADHD.

ELIGIBILITY:
Inclusion Criteria:

* For the proband subjects to be eligible to participate in this study, they need to fit the following criteria: (1) subjects have a clinical diagnosis of ADHD, or Hyperkinetic Disorder defined by the DSM-IV and ICD-10, respectively, which was made by a full-time board-certificated child psychiatrist at the first visit and following visits; (2) their ages range from 6 to 18 when we conduct the study; (3) subjects have at least one biological parent; and (4) both parents are Han Chinese.

Exclusion Criteria:

* The proband subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, Organic Psychosis, or Pervasive Developmental Disorder. Moreover, the subjects will also be excluded from the study if they completely cannot cooperate with blood withdrawal.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects in this study will be recruited from Children's Mental Health Center, Department of Psychiatry, National Taiwan University Hospital (NTUH). The sample will consist of 50 ADHD probands and 50 age- and sex- matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
SNAP-IV | baseline
  self-administered questionnaires to measures ADHD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yung Shang, Ph.D., Principal Investigator — National Taiwan University Hospital